CLINICAL TRIAL: NCT05258747
Title: A Randomized, Open Label, Multi-centre, Two-treatment, Two-period, Two-sequence, Two-stage, Multiple Dose, Steady-state, Crossover, Bioequivalence Study of Olaparib Tablets, 150 mg (Lek Pharmaceuticals d.d.) and Lynparza® (Olaparib) Tablets 150 mg (AstraZeneca Pharmaceuticals LP), in Patients With BRCA Mutated Ovarian Cancer, Recurrent Ovarian Cancer or Metastatic Breast Cancer Under Fasting Condition
Brief Title: A Crossover Bioequivalence Study of Olaparib Tablets, 150 mg (Lek Pharmaceuticals d.d.) and Lynparza® (Olaparib) Tablets 150 mg (AstraZeneca Pharmaceuticals LP), in Patients With Breast Cancer Gene (BRCA) Mutated Ovarian Cancer, Recurrent Ovarian Cancer or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21-VIN-0166/SAN-0647
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: cancer of the ovaries,; female reproductive cancer,; ovarian carcinoma,; female breast cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — olaparib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olaparib tablets, 150 mg, then Lynparza® (olaparib) tablets 150 mg (Other): participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Interventions: Drug: Olaparib tablets, 150 mg; Drug: Lynparza® (olaparib) tablets 150 mg
- Lynparza® (olaparib) tablets 150 mg, then Olaparib tablets, 150 mg (Other): participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Interventions: Drug: Olaparib tablets, 150 mg; Drug: Lynparza® (olaparib) tablets 150 mg

INTERVENTIONS:
Drug: Olaparib tablets, 150 mg — Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia
Drug: Lynparza® (olaparib) tablets 150 mg — Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, Delaware (DE).

SUMMARY:
This is a two-way crossover bioequivalence study between test and reference product in patients diagnosed with BRCA mutated ovarian cancer, recurrent ovarian cancer or metastatic breast cancer.

DETAILED DESCRIPTION:
This is a two-way crossover bioequivalence study between test and reference product in patients diagnosed with BRCA mutated ovarian cancer, recurrent ovarian cancer or metastatic breast cancer.

Patients will be enrolled after providing written informed consent and treatments will be allocated to patient by carrying out randomization using statistical techniques.

Patients that are already on a stable dose of Lynparza® (olaparib) tablets and have met the eligibility criteria will be directly randomized for participation in the study.

After randomization patients will receive either test or reference product in a crossover manner based on the randomization schedule. Patients will receive the dose of 300 mg twice daily for 16 days in a crossover design.

In period-I (Day 1 to Day 8), patients will receive either Test product or Reference product for 8 days based on the randomization schedule.

In period-II (Day 9 to Day 16), patients will be switched to the other product for a second period of 8 days.

ELIGIBILITY:
Inclusion Criteria:

- First-Line Maintenance Treatment of BRCA-mutated Advanced Ovarian Cancer maintenance treatment of adult patients with deleterious or suspected deleterious germline or somatic BRCA-mutated advanced epithelial ovarian, fallopian tube or primary peritoneal cancer who are in complete or partial response to first-line platinum-based chemotherapy.

OR Maintenance Treatment of Recurrent Ovarian Cancer maintenance treatment of adult patients with recurrent epithelial ovarian, fallopian tube or primary peritoneal cancer, who are in complete or partial response to platinum-based chemotherapy.

OR Advanced Germline BRCA-mutated Ovarian Cancer After 3 or More Lines of Chemotherapy treatment of adult patients with deleterious or suspected deleterious germline BRCA-mutated (gBRCAm) advanced ovarian cancer who have been treated with three or more prior lines of chemotherapy.

OR Germline BRCA-mutated Human epidermal growth factor receptor 2 (HER2) -negative Metastatic Breast Cancer treatment of adult patients with deleterious or suspected deleterious gBRCAm, HER2-negative metastatic breast cancer, who have been treated with chemotherapy in the neoadjuvant, adjuvant, or metastatic setting. Patients with hormone receptor (HR)-positive breast cancer should have been treated with a prior endocrine therapy or be considered inappropriate for endocrine therapy.

* Non-smoking, non-pregnant, non-lactating female patient ≥18 years of age with a body mass index (BMI) in the range of 18.50 to 30.00 kg/m^2 (both inclusive).
* Able to give written informed consent for participation in the trial and willing to adhere to protocol requirements.
* Patient having an estimated survival of at least 3 months
* Adequate organ and bone marrow function based upon the following laboratory criteria at the time of eligibility assessment prior to dosing in period 1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Women of non child bearing potential with documented evidence of hysterectomy / bilateral salpingectomy / bilateral oophorectomy at least 6 months prior to Investigational Medicinal Product (IMP) administration or postmenopausal for at least 12 consecutive months.

OR Women of child bearing potential must have negative pregnancy test at screening visit and before randomization and must agree to use an effective method of avoiding pregnancy (including oral, transdermal or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to IMP administration] sexual partner) for at least 4 weeks prior to IMP administration, during the study and up to 6 months after the last dose of IMP. Cessation of birth control after this point should be discussed with a responsible physician.

Exclusion Criteria:

* History of known hypersensitivity to olaparib or its components which, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
* Usage of strong and moderate CYP3A4 inhibitors (e.g., cimetidine, ciprofloxacin, grapefruit juice) or strong and moderate CYP3A4 inducers (e.g., carbamazepine, phenytoin, St. John"s Wort, rifampicin) within 30 days prior to first dosing in Period 01.
* Pregnant or lactating females.
* History or presence of clinically significant lactose, galactose, or fructose intolerance.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (1):
- Sandoz Investigative Site, Vijayawada, Andhra Pradesh, India

RESULTS

PARTICIPANT FLOW:
Groups:
- Olaparib Tablets, 150 mg, Then Lynparza® (Olaparib) Tablets 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, Delaware.
- Lynparza® (Olaparib) Tablets 150 mg, Then Olaparib Tablets, 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, Delaware. Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia
Period: First Period
Arm/Group | Olaparib Tablets, 150 mg, Then Lynparza® (Olaparib) Tablets 150 mg | Lynparza® (Olaparib) Tablets 150 mg, Then Olaparib Tablets, 150 mg
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Second Period
Arm/Group | Olaparib Tablets, 150 mg, Then Lynparza® (Olaparib) Tablets 150 mg | Lynparza® (Olaparib) Tablets 150 mg, Then Olaparib Tablets, 150 mg
Started | 35 | 35
Completed | 34 | 35
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Olaparib Tablets, 150 mg, Then Lynparza® (Olaparib) Tablets 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, DE
- Lynparza® (Olaparib) Tablets 150 mg, Then Olaparib Tablets, 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, DE Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia
- Total: Total of all reporting groups
Arm/Group | Olaparib Tablets, 150 mg, Then Lynparza® (Olaparib) Tablets 150 mg | Lynparza® (Olaparib) Tablets 150 mg, Then Olaparib Tablets, 150 mg | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.77 (8.977) | 50.74 (10.590) | 49.26 (9.859)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 35 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 35 | 35 | 70
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 25.27 (3.480) | 25.62 (3.444) | 25.44 (3.441)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration During the Dosing Interval at Steady State (CmaxSS)
Description: To assess the pharmacokinetics and establish bioequivalence of the Test Product (Olaparib tablets, 150 mg) relative to that of Reference Product (Lynparza® (olaparib) tablets 150 mg) in patients with Breast Cancer Gene (BRCA) mutated ovarian cancer, recurrent ovarian cancer or metastatic breast cancer.
Time Frame: Pre-dose (0.00 hr) on day 1,6,7,8,14,15 and 16 and Post-dose on day 8 and day 16
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Olaparib Tablets, 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia
- Lynparza® (Olaparib) Tablets 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, DE
Arm/Group | Olaparib Tablets, 150 mg | Lynparza® (Olaparib) Tablets 150 mg
Number analyzed (Participants) | 59 | 59
ng/mL | 10395.085 (3374.4800) | 9676.278 (2845.1708)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve for One Dosing Interval at Steady State (AUC(0-t)ss)
Description: To assess the pharmacokinetics and establish bioequivalence of the Test Product (Olaparib tablets, 150 mg) relative to that of Reference Product (Lynparza® (olaparib) tablets 150 mg) in patients with BRCA mutated ovarian cancer, recurrent ovarian cancer or metastatic breast cancer.
Time Frame: Pre-dose (0.00 hr) on day 1,6,7,8,14,15 and 16 and Post-dose on day 8 and day 16
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Olaparib Tablets, 150 mg | Lynparza® (Olaparib) Tablets 150 mg
Number analyzed (Participants) | 59 | 59
hr*ng/mL | 59480.137 (25073.7016) | 64104.218 (29492.0018)

3. Secondary Outcome: Number of Serious Adverse Events
Description: To monitor the serious adverse events of patients and to assess safety of each of the two formulations.
Time Frame: up to Day 24
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Olaparib Tablets, 150 mg | Lynparza® (Olaparib) Tablets 150 mg
Number analyzed (Participants) | 70 | 69
Number of Serious Adverse Events | 0 | 1

4. Secondary Outcome: Number of Adverse Events
Description: To monitor the adverse events of patients and to assess safety of each of the two formulations.
Time Frame: up to Day 24
Measure: Number; unit: Number of Adverse Events
Arm/Group | Olaparib Tablets, 150 mg | Lynparza® (Olaparib) Tablets 150 mg
Number analyzed (Participants) | 70 | 69
Number of Adverse Events | 43 | 37

ADVERSE EVENTS:
Time Frame: From signing informed consent form till end of the study safety assessments (24 days).
Groups:
- Olaparib Tablets, 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, DE
- Lynparza® (Olaparib) Tablets 150 mg: participants will receive 2 x 150 mg Olaparib tablets twice daily for 16 days in a crossover design
  Lynparza® (olaparib) tablets 150 mg: Lynparza® (olaparib) tablets 150 mg Manufactured for: AstraZeneca Pharmaceuticals LP, Wilmington, DE Olaparib tablets, 150 mg: Olaparib tablets, 150 mg of Lek Pharmaceuticals d.d., Slovenia
Arm/Group | Olaparib Tablets, 150 mg | Lynparza® (Olaparib) Tablets 150 mg
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/69
Other Adverse Events (participants affected / at risk) | 19/70 | 17/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib Tablets, 150 mg (N=70) | Lynparza® (Olaparib) Tablets 150 mg (N=69)
Asthenia (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib Tablets, 150 mg (N=70) | Lynparza® (Olaparib) Tablets 150 mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 6 | 4
Asthenia (General disorders) | 4 | 2
White blood cell count decreased (Investigations) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Sandoz's agreements with its investigators may vary. However, Sandoz does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05258747/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT05258747/SAP_001.pdf